CLINICAL TRIAL: NCT03239691
Title: A Phase 2a, Multi-center, Single-blind, Within-subject, Placebo-controlled Study to Assess the Pharmacodynamics of ACT-709478 in Subjects With Photosensitive Epilepsy
Brief Title: A Study to Evaluate the Effect of ACT-709478 in Photosensitive Epilepsy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: AC-083-103
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Photosensitive Epilepsy
MeSH Terms: conditions — Epilepsy, Reflex | interventions — ACT-709478

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-709478 - Single dose administration (Experimental): Up to 16 subjects with photosensitive epilepsy will be studied across a maximum of 4 dose levels. Each dose level will initially be investigated in cohorts of 4 subjects undergoing a fixed sequence of study treatment administration in fed condition
  Interventions: Drug: ACT-709478 for oral use
- Placebo (Placebo Comparator): Placebo will be administered on two study days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-709478 for oral use — Hard gelatin capsules for oral administration formulated at strengths of 10 mg and 100 mg
  Arms: ACT-709478 - Single dose administration
Drug: Placebo — Matching placebo available as matching capsules for oral administration
  Arms: Placebo

SUMMARY:
The main study objective is to assess the effect of ACT-709478 in male and female subjects with photosensitive epilepsy following single dose administration

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure
* Male and female subjects aged between 18 and 60 years (inclusive) at screening
* Photosensitive epilepsy and a generalized PPR in response to IPS of at least 4 units on a SPR in at least 1 condition (eye closure, eyes closed, or eyes open) on 2 occasions at screening with at least 1 hour interval and reproducible on Day -1 (less than 3 units difference in SPR between screening and Day -1)
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use a reliable method of contraception with a failure rate of <1% per year, be sexually inactive, or have a vasectomized partner. Hormonal contraceptives must be initiated at least 1 month before first study treatment administration

Exclusion Criteria:

* Lactating women
* Known hypersensitivity to any of the excipients of the study treatment formulation
* History or clinical evidence of any disease other than epilepsy and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Relevant history of a suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 6 months (categories 4 or 5), or any suicidal behavior within the last 2 years, except for "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), as judged by the investigator using the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening
* History of status epilepticus during the last 12 months
* History of non-epileptic seizures that cannot be differentiated from the participant's epileptic seizures
* History of generalized tonic-clonic seizures triggered by IPS
* Previous history of repeated fainting, syncope, orthostatic hypotension, or vasovagal reactions in the past 5 years
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Individual evaluation of the response to intermittent photic stimulation | From Day 2 to Day 10
  Positive response described as complete suppression of photoparoxysmal response (PPR) or a clinically relevant reduction in the standardized photosensitive range (SPR)

SECONDARY OUTCOMES:
Time to onset of positive response | From Day 2 to Day 10
  Defined by the first time point after ACT-709478 administration at which complete suppression of PPR or clinically relevant reduction in SPR is achieved
Duration of positive response | From Day 2 to Day 10
  Defined as the time elapsed between the time point of onset of the positive response and the last time point of the positive response after ACT-709478 administration
Maximum SPR reduction | From Day 2 to Day 10
  Defined as the largest reduction in SPR achieved at any time point compared to baseline during the positive response after ACT-709478 administration
Time to maximum SPR reduction | From Day 2 to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (5):
- HOSP - Bicêtre Neurologie, Le Kremlin-Bicêtre, France
- Germany (4):
  - Bethel Epilepsy Center, Mara Hospital, Bielefeld
  - Epilepsy Center Frankfurt, Frankfurt
  - Epilepsiezentrum Kork, Kehl
  - Kleinwachau, Sächsisches Epilepsiezentrum Radeberg, Radeberg